CLINICAL TRIAL: NCT06234631
Title: Cannabidiol for Postoperative Opioid Reduction in Primary Total Knee Arthroplasty - a Randomized, Two by Two Factorial, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Cannabidiol for Postoperative Opioid Reduction in Primary Total Knee Arthroplasty
Acronym: CORK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chad Brummett (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Chad Brummett, Professor of Anesthesiology Research, Associate Chair for Research, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00239715; 1U01AR083132-01 (NIH)
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Knee Replacement Surgery; Osteoarthritis, Knee
Keywords: Epidiolex; Pain medication
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized once before surgery and once the day of surgery.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants and the study team at each site will be blinded except for the site research pharmacist and the site project manager (PM) and/or PM delegate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pre - and post-operative CBD (Experimental): Participants will take 300 milligrams (mg)/day on days 1-36 (150mg twice a day [b.i.d.])
  Interventions: Drug: Epidiolex oral solution
- Pre-operative placebo plus post-operative CBD (Experimental): Participants will take placebo prior to surgery days 1-7, then days 8-36 participants will take CBD 300 milligrams (150mg twice a day [b.i.d.])
  Interventions: Drug: Epidiolex oral solution; Other: Placebo
- Pre-operative CBD plus post-operative placebo (Experimental): Participants will take CBD 300 milligrams (mg) /day prior to surgery on days 1-7 (150mg twice a day [b.i.d.]), then days 8-36 will take placebo twice a day [b.i.d.]
  Interventions: Drug: Epidiolex oral solution; Other: Placebo
- Pre- and post-operative placebo (Placebo Comparator): Participants will take placebo on days 1-36 twice a day [b.i.d.]
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Epidiolex oral solution — Participants assigned to CBD will take the medication one hour before or two hours after eating a meal.
  If participants can't tolerate the full-strength dose, the participant can decrease the dosing to 0.75 milliliter twice a day. If this is still not well tolerated, dosing can further be decreased to 0.75 milliliter once per day in the evening.
  Other Names: Cannabidiol
  Arms: Pre - and post-operative CBD; Pre-operative CBD plus post-operative placebo; Pre-operative placebo plus post-operative CBD
Other: Placebo — Participants will be instructed to take one hour before or two hours after eating a meal.
  Arms: Pre- and post-operative placebo; Pre-operative CBD plus post-operative placebo; Pre-operative placebo plus post-operative CBD

SUMMARY:
The goal of this study is to better understand how daily treatment with cannabidiol (CBD) affects the need for opioid pain medication, as well as pain, inflammation and other related symptoms, after knee replacement surgery. The information collected in this study is necessary to help understand whether CBD may be a useful medication before and/or after surgery.

The study hypothesis is that CBD exerts opioid-sparing effects through anti-inflammatory, analgesic, and anxiolytic mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read, understand, and sign the informed consent (English)
* Willingness to participate in all study measures and restrictions, including patient-reported outcomes and longitudinal follow-up
* Scheduled for surgery: primary total knee arthroplasty
* Primary diagnosis of osteoarthritis of the surgical knee
* Individuals of reproductive potential must agree to use acceptable birth control (defined in manual of operating procedures). This includes currently practicing an effective form of two types of birth control for women of childbearing potential, which are defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly from the screening visit until 28 days after the last study drug administration.
* Participants must also agree not to donate sperm or eggs during study drug administration
* Ability to take and to swallow the study medication and be willing to adhere to the treatment regimen
* Agreement to adhere to Lifestyle Considerations (see protocol) throughout study duration

Exclusion Criteria:

* Revision or bilateral total knee arthroplasty
* Individuals receiving or actively applying for worker's compensation or disability and other aspects associated with potential secondary gain
* Severe physical impairment or clinically significant illness (e.g., blindness, paraplegia)
* Co-morbid medical conditions that may significantly impair physical functional status (e.g., current non-skin malignancies, solid organ transplant in the past year)
* Illicit drug use (other than cannabis). Unreported opioid use would be exclusionary but reported prescribed opioid use is allowed (e.g. patient denies opioid use but is found to be positive on the urine drug screen)
* Use of cannabis products in the past 30 days (self-report and confirmed with urinalysis). Note - may be rescreened with appropriate wash-out period (see protocol)
* High daily preoperative opioid dose
* Individuals with major neurological disorders, such as dementia, Parkinson's disease, cognitive impairment, epilepsy, history of traumatic brain injury/head injury, and seizures
* Individuals with significant illness (e.g., cancer) and/or clinically significant labs (e.g. labs measured by complete blood count (CBC) and basic chemistry with values meaningfully outside of the normal range [abnormal levels to be reviewed by the Principal Investigator or prescribing provider])
* Medical or psychiatric conditions that in the judgment of study personnel would preclude participation in this study (e.g., psychosis, suicidal ideation; note that stable anxiety and depression are not exclusions)
* Pregnant or nursing women (total joint arthroplasty is typically not indicated in this group of patients)
* Self-reported liver cirrhosis
* Self-reported uncontrolled diabetes
* Self-reported active hepatitis (any etiology, including infectious, autoimmune, or alcohol-related)
* Blood pressure at screening above 180 millimeters of mercury (mmHg) systolic and/or 120 mmHg diastolic; if value exceeds the set point, potential participants will have repeat assessment within 5 minutes for up to two additional measurements.
* Resting heart rate at screening less than 50 beats per minute (bpm) or greater than 100 bpm; if value exceeds the set point, potential participants will have repeat assessment within 5 minutes for up to two additional measurements.
* Elevated liver enzymes and bilirubin (measured by blood test at screening)
* Serum total bilirubin ≥ 2.5 milligrams (mg) per deciliter (dL) (mg/dL); or,

  * Alanine transaminase (ALT) or Alanine transaminase (AST) ≥ 3x upper limit normal (ULN); or,
  * Alkaline phosphatase ≥ 2x ULN
* Severe cardiovascular disease (e.g., current unstable angina, current congestive heart failure, or current severe valvular abnormalities) that is self-reported by patient or in medical record
* Current valproate, clobazam, or warfarin use per self-report or medical records
* Current use of strong inducers of cytochrome p450 (CYP) enzymes CYP3A4 and CYP2C19, or CYP2C19 substrates with a narrow therapeutic index
* Self-reported allergies to sesame oil, strawberries, opioids, or cannabis/cannabinoids
* Any impairment, activity, behavior, or situation that in the judgment of the study team would prevent satisfactory completion of the study protocol
* Self-reported severe side effects to opioids precluding the use of opioids for post-surgical pain and/or clear plan not to use any opioids after surgery
* Participation in other clinical trials over the course of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Total postoperative opioid consumption (measured in oral morphine equivalents) during the 28 days after surgery | 28 days (after surgery)

SECONDARY OUTCOMES:
The number of treatment-emergent adverse events (TEAEs) | Five weeks of study treatment (Days 1 - 36)
Proportion of participants with at least one treatment-emergent adverse events (TEAEs) | Five weeks of study treatment (Days 1 - 36)
The Number of serious adverse events (SAEs) | Five weeks of study treatment (Days 1 - 36)
Proportion of participants with at least one serious adverse event (SAE) | Five weeks of study treatment (Days 1 - 36)
Number of deaths due to any cause | Five weeks of study treatment (Days 1 - 36)
Frequency of deaths due to any cause | Five weeks of study treatment (Days 1 - 36)
Proportion of participants that prematurely discontinue study medications because of TEAE | Five weeks of study treatment (Days 1 - 36)
Percentage of participants that meet or exceed the thresholds of liver enzymes | Five weeks of study treatment (Days 1 - 36)
  Protocol eligibility exclusion includes:
  * Serum total bilirubin ≥ 2.5 milligrams (mg) per deciliter (dL) (mg/dL)
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3x upper limit normal (ULN)
  * Alkaline phosphatase ≥ 2x ULN
Total postoperative opioid consumption (measured in oral morphine equivalents (OME)) during the 28 days after surgery and the pre-operative phase | 36 days (pre-post operative)
  This is the same outcome as the primary outcome but this secondary endpoint will address the effect of pre-operatively administered CBD and Placebo.
Worst pain intensity for surgical site between groups during 7-day epochs from day of surgery through end of active intervention | Days 8-36 (post-surgery)
  This is a scale from 0-10 (numerical rating scale, 10 worse pain) in which the participants rate the worse pain.
Anxiety based on the Patient-Reported Outcomes Measurement Information System (PROMIS)-29+2 profile v2.1 | pre-op days 1-7
  There are 4-questions on this survey regarding anxiety. Participants answer the questions from never (1) to always (5). Scores range from 4-20 with a higher score indicating higher levels of anxiety.
Anxiety based on the Patient-Reported Outcomes Measurement Information System (PROMIS)-29+2 profile v2.1 | post-op days 8-36
  There are 4-questions on this survey regarding anxiety. Participants answer the questions from never (1) to always (5). Scores range from 4-20 with a higher score indicating higher levels of anxiety.
Sleep disturbance on the PROMIS-29+2 v.2.1 | pre-op days 1-7
  There are 4-questions on this survey regarding sleep disturbance with a likert type scale.
  Scores range from 4-20 with a higher score indicating higher levels of sleep disturbance.
Sleep disturbance on the PROMIS-29+2 v.2.1 | post-op days 8-36
  There are 4-questions on this survey regarding sleep disturbance with a likert type scale.
  Scores range from 4-20 with a higher score indicating higher levels of sleep disturbance.
Change in Interleukin-6 (IL-6) levels in the blood (University of michigan site only) | Baseline, up to day 36 (post -surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Brummett, MD, Principal Investigator — University of Michigan; Kevin F Boehnke, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
The final de-identified, anonymized dataset or the minimum necessary will be available upon request or from a University of Michigan repository. The final dataset will include demographics, perioperative medical record data, patient-reported outcomes, daily pain and medication diary data, functional testing scores, and biomarkers of inflammation and pharmacokinetics. The study team anticipates 1 data file with baseline, day of surgery, 2 week, 1-month, 3-month, and 6-month follow-up data.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available by request 5 years after the completion of the primary endpoint.
Access Criteria: Access may be requested by contacting PI, Dr. Chad Brummett at cbrummet@umich.edu or the University of Michigan repository. A data use agreement may also be required.